CLINICAL TRIAL: NCT06810752
Title: Thyme Honey for Management of Oral Lichen Planus: A Non- Inferiority Controlled Randomized Clinical Trial
Brief Title: Thyme Honey for Management of Oral Lichen Planus
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-092
Record Dates: First submitted 2025-01-23; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-10

CONDITIONS: Oral Lichen Planus
Keywords: Oral Lichen Planus; Thyme Honey; triamcinolone acteonide
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Thyme Honey group (Active Comparator): Topical application of Thyme Honey
  Interventions: Dietary Supplement: thyme honey
- Control group (Placebo Comparator): Topical application of Triamcinolone acetonide
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Dietary Supplement: thyme honey — Topical application on the oral mucosa
  Arms: Thyme Honey group
Drug: Triamcinolone Acetonide — Topical application on the oral mucosa
  Arms: Control group

SUMMARY:
the study aimed to assess the effect of topical application of thyme honey in comparison to 0.1% triamcinolone acetonide oral paste on the relief of pain and clinical improvement in patients with OLP

ELIGIBILITY:
Inclusion Criteria:• Patients clinically and histopathologically (if required) diagnosed as suffering from OLP.

* Patients free from any visible oral lesions other than OLP.
* Patients who agreed to take supplied medications.
* Patients who agreed for the biopsy (when required).

Exclusion Criteria:• •Patients suffering from any systemic disease.

* Treatment with any systemic treatment such as systemic steroids, other immunosuppressive drugs or non-steroidal anti-inflammatory drugs at least eight weeks.
* Treatment with any oral topical medications for at least four weeks prior to the study.
* Pregnant and lactating women.
* In addition, no consideration was given to patients with a history of hypersensitivity to honey.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
VAS score assessement | 1 month
  Pain intensity

SECONDARY OUTCOMES:
measurement of salivary level of miRna155 | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- The British university in Egypt, Cairo, Egypt